CLINICAL TRIAL: NCT03389737
Title: The Effects of the Novel "Step Up Your Game" Program on Men's Collegiate Lacrosse Players: A Comparative Study of a Comprehensive Osteopathic Approach on Performance
Brief Title: The Effects of the Novel "Step Up Your Game" Program on Men's Lacrosse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Hallie Zwibel, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BHS-1261
Record Dates: First submitted 2017-12-20; First posted 2018-01-04 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental group will have monthly contact with the physicians, during which the athletes will receive individualized care and guidance in support of their performance goals.
  Interventions: Behavioral: Counseling
- Control (Active Comparator): Control group will not have monthly contact with the physicians.
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Counseling on healthy behaviors with in person meetings.
  Arms: Experimental
Behavioral: Counseling — Counseling on healthy behaviors with emails.
  Arms: Control

SUMMARY:
For the purpose of this pilot study, the investigators hypothesize that the use of the Step Up Your Game protocol will result in statistically significant improvements in health and athletic performance. The key to this is the coordination of resources from a supervising physician, physical therapist, trainer, dietitian, coach, competitor, role model, psychologist, and spiritual leader. Notably, Step Up Your Game provides resources which would allow patients to find or be their own physical therapist, trainer, dietitian, coach, competitor, role model, psychologist, and spiritual leader. The role of the supervising physician, however, is meant for a qualified professional, who follows the osteopathic approach to medicine, in which the body is treated as an integrated whole, while also working to prevent and treat injuries. Though not limited solely to osteopathic physicians, it is critical to take into account every health aim and injury in the context of the athlete and how these affect all aspects of participants lives.

ELIGIBILITY:
Inclusion Criteria:

* Individuals capable of giving consent between ages of 18 and 22.
* Must be members of the NYIT lacrosse team.

Exclusion Criteria:

* Individuals who are not able to participate throughout the season whether it's due to a medical problem or academic probation.
* Individuals who are receiving sports related medical care other than that from the physician in study.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men's Lacrosse team at NYIT
Enrollment: 25 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
RAND-36 Survey | 3 months
  Short form health survey

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 | 3 months
  Depression scale. Indicates depression severity with higher scores meaning more severe depression.
Lean muscle mass | 3 months
  Percent lean muscle mass
Adipose tissue | 3 months
  Percent adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Hallie Zwibel, D.O., Principal Investigator — NYIT
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers may contact PI for details.
Supporting Information: Study Protocol
Time Frame: 1 year